CLINICAL TRIAL: NCT00316108
Title: Boston Scientific EPI: A Carotid Stenting Trial for High-Risk Surgical Patients
Brief Title: Boston Scientific Embolic Protection, Inc. (EPI): A Carotid Stenting Trial for High-Risk Surgical Patients (BEACH)
Acronym: BEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S5385; COR2000001U
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Carotid Artery Diseases; Stroke; Cerebral Arteriosclerosis
Keywords: Carotid; Carotid Artery Stenting; Stent; Carotid Endarterectomy; Stroke; Transient Ischemic Attack; Stenosis; Atherosclerotic Disease
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Intracranial Arteriosclerosis; Ischemic Attack, Transient; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Device: WALLSTENT® Endoprosthesis™

INTERVENTIONS:
Device: WALLSTENT® Endoprosthesis™ — Carotid Artery Stent

SUMMARY:
The purpose of this study is to determine whether morbidity and mortality for high-risk surgical patients treated with the Carotid Wallstent in conjunction with the FilterWire EX and EZ System distal protection device will be less than or equal to that of objective performance criteria (OPC) derived from historic controls undergoing surgical intervention with a carotid endarterectomy (CEA).

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in this country with approximately 600,000 new stroke cases each year. Mortality rates as high as 40 percent have been reported for stroke as a result of ischemia associated with the carotid distribution. Currently, the primary therapy for carotid artery occlusive disease is carotid endarterectomy (CEA) or the surgical removal of atheromatous material from inside the artery.

Although CEA is an effective treatment for the majority of patients with carotid occlusive disease, there remains a need for a treatment option for those patients with significant surgical risk factors. These patients have been shown to have much higher rates of morbidity and mortality. There are approximately 50,000-70,000 patients each year who are considered poor surgical candidates. These patients present with either one or more anatomical or co-morbid conditions and have a one-year stroke and death rate of up to 15% with traditional surgical treatment.

Carotid artery stenting (CAS) has been reported by numerous single-center trials to be feasible in the treatment of carotid artery stenosis. Moreover, the risk benefit ratio has been suggested to be the largest in those patients with a higher risk profile for the CEA treatment option.

This trial will study the effects of percutaneous intervention using the Monorail™ Carotid Wallstent® Endoprosthesis (Carotid Wallstent) in conjunction with the FilterWire System distal protection device (FilterWire EX and EZ) on rates of common peri-procedural complications as well as on long-term outcomes as compared to historical outcomes of patients undergoing CEA.

ELIGIBILITY:
Key General Inclusion Criteria:

* Patient must meet criteria for either A or B:

A. Symptomatic: Carotid stenosis of greater than or equal to 50% via angiography with associated cerebral or retinal TIA or ischemic stroke symptoms within 180 days of the procedure, which are determined to have occurred in the cerebral hemisphere or eye ipsilateral to the target carotid artery lesion and to be reasonably attributable to that lesion; or

B. Asymptomatic: Carotid stenosis greater than or equal to 80% via angiography without associated cerebral or retinal TIA or ischemic stroke symptoms within 180 days of the procedure.

* Target lesion is in the native common carotid artery (CCA), internal carotid artery (ICA), or carotid bifurcation.
* Target arterial segment to be stented has a diameter of greater than or equal to 4.0 mm to less than or equal to 9.0 mm.
* Vessel diameter distal to the target lesion is greater than or equal to 3.5 mm and less than or equal to 5.5 mm as an optimal "landing zone" for placement of the FilterWire EZ System with visual angiographic recommendations as described in the instructions for use (IFU).

Key High-Risk Eligibility Inclusion Criteria:

* Patients must qualify in at least one high-risk category. The high-risk categories are defined as:

  * Anatomical conditions [one (1) criterion qualifies]
  * Co-morbid conditions Class I [one (1) criterion qualifies]
  * Co-morbid conditions Class II [two (2) criteria qualify]

Exclusion Criteria:

* Patient has experienced an evolving, acute, or recent stroke within 21 days of study evaluation.
* A total occlusion of the ipsilateral carotid artery. (Only for Roll-In and Pivotal patients.)
* A total occlusion of the contralateral carotid artery. (Only for Bilateral Registry patients.)
* Pre-existing stent(s):

  * Roll-In and Pivotal Patients: located within the ipsilateral carotid distribution; a stent was placed in a contralateral vessel within the previous 30 days of the study enrollment.
  * Bilateral Registry Patients: located within the carotid distribution.
* A target lesion which is expected to require more than one stent.
* Known cardiac sources of emboli of a type likely to be associated with cerebral ischemic events [e.g. endocarditis, intracardiac thrombus, embolic-associated cardiovascular lesions, or any current arrhythmia (e.g. atrial fibrillation, atrial flutter, etc.)].
* Myocardial infarction (MI) within 72 hours prior to the index procedure, defined as creatine kinase (CK)-MB > 2 X the local laboratory's upper limit of normal (ULN).
* Any surgery requiring general anesthesia (e.g. coronary artery bypass graft [CABG], valve replacement, or abdominal aortic aneurysm) less than or equal to 30 days preceding the stent procedure.
* The patient is enrolled in another investigational study protocol and has not completed the required follow-up period of the evaluation. The patient may not participate in another investigational study that may confound the treatment or outcomes of the BEACH protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2002-02; Primary Completion 2005-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is one-year morbidity and mortality, defined as the cumulative incidence of any non Q-wave myocardial infarction within the 24 hours following carotid stenting | 1 year
peri-procedural (within 30 days of procedure) death, stroke, Q-wave myocardial infarction | Within 30 days of Procedure
late ipsilateral stroke or death due to neurologic events from 31 days up to and including twelve-month follow-up. | 1 year

SECONDARY OUTCOMES:
Peri-procedural morbidity and mortality | Within 30 Days of procedure
FilterWire EX and EZ System technical success | Post procedure
Carotid Wallstent technical success | Post Procedure
system technical success | Post Procedure
angiographic success | Post Procedure
procedural success | Post Procedure
30-day clinical success | 30 days post procedure
peri-procedural overall morbidity | 30 days post procedure
one-year clinical success | 1 Year post procedure
late stroke, transient ischemic attack (TIA) and death. | 1 year post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher White, MD, Principal Investigator — Ochsner Health System; Sriram Iyer, MD, Principal Investigator — Lenox Hill Heart and Vascular Institute; Pamela G Grady, Ph.D, Study Director — Boston Scientific Corporation
Locations (50):
- United States (50):
  - Bapatist Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital, Newport Beach, California
  - St. Joseph's Medical Center, Stockton, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami School of Medicine - Jackson Memorial Hospital, Miami, Florida
  - Miami Cardiac and Vascular Institute, Miami, Florida
  - Northwest Medical Center, Plantation, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - St. Joseph's Hospital of Atlanta/American Cardiovascular Research Institute, Atlanta, Georgia
  - Rush Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - St. Francis Medical Center, Peoria, Illinois
  - St. John's Hospital - Prairie Heart Institute, Springfield, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Wayne State University- Detroit Medical Center, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kaleida Health/Millard Fillmore Hospital, Buffalo, New York
  - Lenox Hill Heart and Vascular Institute, New York, New York
  - New York Presbyterian Hospital/Columbia Vascular Interventional Radiology, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic & Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Hahnemann University/ Tenet Healthcare Corporation, Philadelphia, Pennsylvania
  - UPMC-Shadyside Hospital Pittsburgh Vascular Institute, Pittsburgh, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - Providence Hospital South Carolina Heart Center, Columbia, South Carolina
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Skyline Medical Center/ Howell Allen Clinic, Nashville, Tennessee
  - St. Luke's Episcopal Hospital Texas Heart Institute, Houston, Texas
  - University of Texas-Houston Medical School, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Baptist Hospital, San Antonio, Texas
  - LDS Hospital, Salt Lake City, Utah
  - St. Mary's Hospital, Richmond, Virginia
  - Deaconess Medical Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Iyer SS, White CJ, Hopkins LN, Katzen BT, Safian R, Wholey MH, Gray WA, Ciocca R, Bachinsky WB, Ansel G, Joye JD, Russell ME; BEACH Investigators. Carotid artery revascularization in high-surgical-risk patients using the Carotid WALLSTENT and FilterWire EX/EZ: 1-year outcomes in the BEACH Pivotal Group. J Am Coll Cardiol. 2008 Jan 29;51(4):427-34. doi: 10.1016/j.jacc.2007.09.045. PMID 18222352